CLINICAL TRIAL: NCT00926536
Title: Impact of C-arm CT in Patients With Hepatocellular Carcinoma (HCC) Undergoing Transhepatic Arterial Chemoembolization (TACE): Optimal Imaging Guidance
Brief Title: Impact of C-arm CT in Patients With HCC Undergoing TACE: Optimal Imaging Guidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Siemens Healthcare Diagnostics Inc (Industry)
Responsible Party: Principal Investigator, Nishita Kothary, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-15849; SU-05122009-2518 (Other: Stanford University); HEP0020 (Other: OnCore)
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C-arm CT + DSA as needed' (Experimental): In the group of subjects randomized in this group, the image guidance component of the procedure will be conducted by the acquisition of 3D CT-like images during a trans-hepatic arterial injection of iodinated contrast agent for road mapping the tumor feeding vessels and supplemented by DSA as needed by the operating physician as imaging guidance for planning tumor(s) treatment approach.
  Interventions: Device: C-arm CT + DSA as needed
- DSA only (Active Comparator): In the group of subjects randomized in this group, present standard of care, i.e DSA imaging only will be used by the operating physician to map out the tumor vessels and used for treatment approach. Additional 3D CT-like images will be obtained, but only used if the operator cannot perform adequate planning using DSA alone.
  Interventions: Device: DSA only

INTERVENTIONS:
Device: C-arm CT + DSA as needed — C-arm CT images obtained and supplemented with DSA if needed
  Other Names: x-ray image intensifier; C-arm CT
  Arms: C-arm CT + DSA as needed'
Device: DSA only — DSA imaging only
  Other Names: Standard of care
  Arms: DSA only

SUMMARY:
Patients will be enrolled based on presence of HCC and eligibility for TACE. They will be randomized to one of two arms for imaging navigation to the optimal catheter location for chemotherapy injection to treat the first (possibly sole) tumor target. The two arms will be: TACE using C-arm CT supplemented by DSA or DSA only (only DSA images will be used for navigation and tumor vessel tracking). Navigation to subsequent treatment targets in all patients will be done with fluoroscopy, CACT, and DSA, as is standard of care at Stanford University Medical Center, and is not part of the study. Vascular complexity, which affects navigation difficulty and thus the need for imaging, will be assessed separately for use in data analysis by two radiologists on a four-point scale.

DETAILED DESCRIPTION:
We hope to learn more about the utility of C-arm CT in patients undergoing TACE for HCC. Data will be evaluated with regards to:

1. Sensitivity and specificity to diagnose additional tumors and its impact on transplantation criteria.
2. The ability to decrease procedural time by aiding navigation through complex arterial anatomy.
3. Impact on radiation dose. Although the patient would receive the radiation during C-arm CT, overall the number of DSA angiograms and fluroscopy may decrease, potentially negating any effect of the additional dose from C-arm CT

ELIGIBILITY:
Inclusion Criteria:

Patients must be affected by HCC

Patients must be 18 years old or older

Patients must have received an abdominal CT, PET/CT scan or MRI, completed prior to the TACE procedure.

Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Subjects under the age of 18

Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rebecca Fahrig, Principal Investigator — Stanford University; Nishita N. Kothary, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was open from 01/13/2009 thru 10/13/2010. During this period, subjects with HCC who were scheduled to undergo TACE were approached for permission to participate in the study.
Groups:
- C-arm CT +DSA as Needed: C-arm CT in imaging guidance of TACE supplemented with DSA as needed for vessel tracking and navigation
- DSA Only: Only Digital subtraction images used for vessel tracking and tumor navigation
Period: Overall Study
Arm/Group | C-arm CT +DSA as Needed | DSA Only
Started | 44 | 43
Completed | 43 | 41
Not Completed | 1 | 2
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Population: Only patients completing the study are represented here. The three patients that were excluded by the physician is because the patients disease had progressed by the time of the study
Groups:
- C-arm CT + DSA as Needed: C-arm CT in imaging guidance of TACE supplemented by DSA as needed for vessel navigation and tracking
- DSA Only: DSA images only used for vessel navigation and tracking
- Total: Total of all reporting groups
Arm/Group | C-arm CT + DSA as Needed | DSA Only | Total
Number analyzed (Participants) | 43 | 41 | 84
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Over 18 years old | 43 | 41 | 84
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18
  Male | 37 | 29 | 66

OUTCOME MEASURES:

1. Primary Outcome: Dose Area Product (DAP)
Description: Dose area product (DAP) is a measure of the entire amount of energy (radiation dose) delivered to the patient by the beam (indicator of stochastic dose)
Time Frame: Duration of a TACE procedure, an average of 2 hours
Population: DAP measured in both groups
Measure: Mean (Full Range); unit: Gy.cm2
Groups:
- C-arm CT +DSA as Needed: C-arm CT images used for navigational purposes supplemented by DSA if needed
- DSA Only: Only DSA imaging used for navigational purposes
Arm/Group | C-arm CT +DSA as Needed | DSA Only
Number analyzed (Participants) | 43 | 41
Gy.cm2 | 184.2 [148.2 to 220.2] | 137.4 [101.1 to 173.7]
Statistical Analysis 1: Comparison: C-arm CT +DSA as Needed vs DSA Only; Test type: Superiority or Other; p < .001, Mixed Models Analysis — Decrease in DAP in C-arm CT +DSA group when compared to DSA only; Mean Difference (Net) = 71.6

2. Primary Outcome: Cumulative Dose (CD), a Measure of Radiation Dose
Description: CD - a measurement of total radiation to the skin (measure of a deterministic dose)
Time Frame: Duration of a TACE procedure, an average of 2 hours
Population: CD measured in both groups
Measure: Mean (Full Range); unit: mGy
Arm/Group | C-arm CT +DSA as Needed | DSA Only
Number analyzed (Participants) | 43 | 41
mGy | 626.4 [439.5 to 813.3] | 784.7 [537.3 to 1032.1]
Statistical Analysis 1: Comparison: C-arm CT +DSA as Needed vs DSA Only; Test type: Superiority or Other; p = 0.017, Mixed Models Analysis — Decrease in CD in C-arm CT +DSA group when compared to DSA only; Mean Difference (Net) = 158.3

ADVERSE EVENTS:
Time Frame: The duration of the procedure, since this was an imaging study. TACE procedures are an average of 2 hours.
Groups:
- C-arm CT + DSA as Needed: C-arm CT used for the purposes of navigation, supplemented by DSA if needed
- DSA Only: DSA only used for navigation
Arm/Group | C-arm CT + DSA as Needed | DSA Only
Serious Adverse Events (participants affected / at risk) | 0/43 | 1/41
Other Adverse Events (participants affected / at risk) | 0/43 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C-arm CT + DSA as Needed (N=43) | DSA Only (N=41)
Arterial Hematoma (Surgical and medical procedures) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This is an imaging study looking at two different modalities of imaging. There is no long term follow up or A/Es associated with this type of a study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less